CLINICAL TRIAL: NCT04665050
Title: A Phase 1, Randomized, Double-blind, Active-Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Polyvalent Pneumococcal Conjugate Vaccine in Healthy Japanese Adults.
Brief Title: Safety, Tolerability, and Immunogenicity of a Polyvalent Pneumococcal Conjugate Vaccine (V116) in Japanese Adults (V116-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: pPCV-002; pPCV-002 (Other: Merck); jRCT2071200094 (Registry Identifier: jRCT); V116-002 (Other: Merck)
Record Dates: First submitted 2020-12-08; First posted 2020-12-11 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V116 (Experimental): Participants receive a single 1.0 mL intramuscular (IM) injection of V116 on Day 1.
  Interventions: Biological: V116
- PNEUMOVAX™23 (Active Comparator): Participants receive a single 0.5 mL IM injection of PNEUMOVAX™23 on Day 1.
  Interventions: Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 2 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Polyvalent pneumococcal conjugate vaccine (pPCV); Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116
Biological: PNEUMOVAX™23 — Pneumococcal 23-valent polyvalent vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PPSV23
  Arms: PNEUMOVAX™23

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and immunogenicity of a polyvalent pneumococcal conjugate vaccine (V116) with that of PNEUMOVAX™23 in healthy Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

* is a healthy Japanese male or female ≥20 years of age at time of randomization
* male participants must agree to be abstinent or use contraception during the intervention period and for ≥30 days after the last dose of study intervention
* female participants must not be pregnant or breastfeeding, and is either:
* not a woman of childbearing potential (WOCBP) or
* a WOCBP who agrees to remain abstinent or use contraception during the intervention period and for ≥30 days after the last dose of study intervention

Exclusion Criteria:

* has a history of invasive pneumococcal disease (IPD) within 3 years of Day 1
* has a known hypersensitivity to any vaccine components
* has impaired immunological function
* has a coagulation disorder
* had a recent febrile illness (axillary temperature ≥37.5°C or equivalent) within 72 hours before Day 1
* has a known malignancy that is progressing/requiring treatment
* has received, or is expected to receive, a pneumococcal vaccine outside the study protocol
* has received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed the regimen for ≥30 days prior to Day 1
* is receiving immunosuppressive therapy
* has received any non-live vaccine from 14 days prior to Day 1 other than inactivated influenza vaccine
* has received any live vaccine from 30 days prior to Day 1
* has received a blood transfusion or blood products
* has participated in another clinical trial within 2 months of this study
* has clinically relevant drug or alcohol abuse
* has any condition that, in the opinion of the investigator, precludes participation in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Japan (2):
  - Souseikai PS Clinic ( Site 0201), Fukuoka
  - Souseikai Nishikumamoto Hospital ( Site 0202), Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Haranaka M, Yono M, Kishino H, Igarashi R, Oshima N, Sawata M, Platt HL. Safety, tolerability, and immunogenicity of a 21-valent pneumococcal conjugate vaccine, V116, in Japanese healthy adults: A Phase I study. Hum Vaccin Immunother. 2023 Aug 1;19(2):2228162. doi: 10.1080/21645515.2023.2228162. PMID 37389808

RESULTS

PARTICIPANT FLOW:
Groups:
- V116: Participants received a single 1.0 mL intramuscular (IM) injection of V116 on Day 1.
- PNEUMOVAX™23: Participants received a single 0.5 mL IM injection of PNEUMOVAX™23 on Day 1.
Period: Overall Study
Arm/Group | V116 | PNEUMOVAX™23
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V116 | PNEUMOVAX™23 | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (13.7) | 64.0 (12.7) | 63.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 51 | 51 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs included tenderness/pain, redness/erythema, and swelling. The percentage of participants with one or more solicited injection-site AE was reported for each arm.
Time Frame: Up to 5 days postvaccination
Population: All randomized participants who received study vaccination
Measure: Number; unit: Percentage of Participants
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Percentage of Participants
  Injection site erythema | 9.8 | 9.8
  Injection site pain | 54.9 | 66.7
  Injection site swelling | 13.7 | 13.7
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Injection Site Erythema; Test type: Other — Estimated difference and confidence interval (CI) are calculated based on the Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-12.7 to 12.7] — V116 minus PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Injection Site Pain; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = -11.8, 95% CI 2-sided [-30.0 to 7.3] — V116 minus PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Injection Site Swelling; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-14.1 to 14.1] — V116 minus PNEUMOVAX™23

2. Primary Outcome: Percentage of Participants With a Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs included headache, muscle pain/myalgia, joint pain/arthralgia, and tiredness/fatigue. The percentage of participants with one or more solicited systemic AE was reported for each arm.
Time Frame: Up to 5 days postvaccination
Population: All randomized participants who received study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Percentage of participants
  Fatigue | 13.7 | 9.8
  Arthralgia | 3.9 | 3.9
  Myalgia | 17.6 | 19.6
  Headache | 9.8 | 9.8
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Fatigue; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = 3.9, 95% CI 2-sided [-9.4 to 17.5] — V116 minus PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Arthralgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-9.9 to 9.9] — V116 minus PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Myalgia; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = -2.0, 95% CI 2-sided [-17.5 to 13.6] — V116 minus PNEUMOVAX™23
Statistical Analysis 4: Comparison: V116 vs PNEUMOVAX™23; Headache; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-12.7 to 12.7] — V116 minus PNEUMOVAX™23

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE)
Description: An SAE is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. SAEs that were reported by the investigator to be at least possibly related to the study vaccination were reported.
Time Frame: Up to 62 days postvaccination
Population: All randomized participants who received study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Percentage of participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Test type: Other — Estimated difference and CI are calculated based on the Miettinen & Nurminen method; Difference in percentage = 0.0, 95% CI 2-sided [-7.1 to 7.1] — V116 minus PNEUMOVAX™23

4. Secondary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the Common Serotypes in V116 and PNEUMOVAX™23
Description: The serotype-specific OPA GMTs for serotypes common to V116 and PNEUMOVAX™23 were determined using the multiplex opsonophagocytic assay (MOPA). Serotype-specific OPA GMTs and GMT ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) model. Per protocol, within-group measures of dispersion (MOD) were not calculated.
Time Frame: Day 30 postvaccination
Population: All randomized participants without deviations from the protocol that may have substantially affected the results of this immunogenicity endpoint and who had sufficient data to perform the analyses
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Titers
  Serotype 3 | 161.08 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 100.76 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 5327.67 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4406.11 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 1479.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 738.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 5768.79 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3000.50 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 33187.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 28831.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 1287.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 721.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 6555.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3466.72 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 3608.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1330.75 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 1467.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 603.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 1356.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 563.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 8470.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3293.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 3542.90 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1553.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Serotype 3; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.60, 95% CI 2-sided [1.07 to 2.40] — V116/PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Serotype 7F; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.21, 95% CI 2-sided [0.69 to 2.11] — V116/PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Serotype 19A; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.00, 95% CI 2-sided [1.24 to 3.24] — V116/PNEUMOVAX™23
Statistical Analysis 4: Comparison: V116 vs PNEUMOVAX™23; Serotype 22F; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.92, 95% CI 2-sided [1.04 to 3.57] — V116/PNEUMOVAX™23
Statistical Analysis 5: Comparison: V116 vs PNEUMOVAX™23; Serotype 33F; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.15, 95% CI 2-sided [0.71 to 1.86] — V116/PNEUMOVAX™23
Statistical Analysis 6: Comparison: V116 vs PNEUMOVAX™23; Serotype 8; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.78, 95% CI 2-sided [1.24 to 2.58] — V116/PNEUMOVAX™23
Statistical Analysis 7: Comparison: V116 vs PNEUMOVAX™23; Serotype 9N; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 1.89, 95% CI 2-sided [1.19 to 3.00] — V116/PNEUMOVAX™23
Statistical Analysis 8: Comparison: V116 vs PNEUMOVAX™23; Serotype 10A; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.71, 95% CI 2-sided [1.47 to 5.00] — V116/PNEUMOVAX™23
Statistical Analysis 9: Comparison: V116 vs PNEUMOVAX™23; Serotype 11A; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.43, 95% CI 2-sided [1.52 to 3.89] — V116/PNEUMOVAX™23
Statistical Analysis 10: Comparison: V116 vs PNEUMOVAX™23; Serotype 12F; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.40, 95% CI 2-sided [1.20 to 4.83] — V116/PNEUMOVAX™23
Statistical Analysis 11: Comparison: V116 vs PNEUMOVAX™23; Serotype 17F; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.57, 95% CI 2-sided [1.59 to 4.17] — V116/PNEUMOVAX™23
Statistical Analysis 12: Comparison: V116 vs PNEUMOVAX™23; Serotype 20A; Test type: Other — GMT ratio and 95% confidence interval CI are estimated from a cLDA model; GMT Ratio = 2.28, 95% CI 2-sided [1.46 to 3.56] — V116/PNEUMOVAX™23

5. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the Common Serotypes in V116 and PNEUMOVAX™23
Description: The GMCs for serotype-specific pneumococcal IgG antibodies were measured using pneumococcal electrochemiluminescence (PnECL). Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% CIs were calculated using a cLDA model. Per protocol, within-group MOD were not calculated.
Time Frame: Day 30 postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
μg/mL
  Serotype 3 | 1.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.73 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F | 10.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A | 10.75 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F | 3.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.69 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F | 22.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 14.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8 | 19.38 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N | 14.17 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A | 11.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A | 9.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F | 2.87 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F | 19.46 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A | 23.53 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11.46 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Serotype 3; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.54, 95% CI 2-sided [1.08 to 2.21] — V116/PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Serotype 7F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.21, 95% CI 2-sided [1.36 to 3.60] — V116/PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Serotype 19A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.16, 95% CI 2-sided [1.45 to 3.23] — V116/PNEUMOVAX™23
Statistical Analysis 4: Comparison: V116 vs PNEUMOVAX™23; Serotype 22F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.33, 95% CI 2-sided [1.36 to 3.99] — V116/PNEUMOVAX™23
Statistical Analysis 5: Comparison: V116 vs PNEUMOVAX™23; Serotype 33F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.52, 95% CI 2-sided [0.97 to 2.37] — V116/PNEUMOVAX™23
Statistical Analysis 6: Comparison: V116 vs PNEUMOVAX™23; Serotype 8; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.88, 95% CI 2-sided [1.32 to 2.68] — V116/PNEUMOVAX™23
Statistical Analysis 7: Comparison: V116 vs PNEUMOVAX™23; Serotype 9N; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.37, 95% CI 2-sided [1.49 to 3.74] — V116/PNEUMOVAX™23
Statistical Analysis 8: Comparison: V116 vs PNEUMOVAX™23; Serotype 10A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.16, 95% CI 2-sided [1.28 to 3.65] — V116/PNEUMOVAX™23
Statistical Analysis 9: Comparison: V116 vs PNEUMOVAX™23; Serotype 11A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.92, 95% CI 2-sided [1.28 to 2.89] — V116/PNEUMOVAX™23
Statistical Analysis 10: Comparison: V116 vs PNEUMOVAX™23; Serotype 12F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 3.49, 95% CI 2-sided [1.94 to 6.27] — V116/PNEUMOVAX™23
Statistical Analysis 11: Comparison: V116 vs PNEUMOVAX™23; Serotype 17F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.88, 95% CI 2-sided [1.92 to 4.31] — V116/PNEUMOVAX™23
Statistical Analysis 12: Comparison: V116 vs PNEUMOVAX™23; Serotype 20A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 2.05, 95% CI 2-sided [1.30 to 3.25] — V116/PNEUMOVAX™23

6. Secondary Outcome: Serotype-specific OPA GMTs for the Unique Serotypes in V116
Description: The serotype-specific OPA GMTs for serotypes unique to V116 were determined using the MOPA. Serotype-specific OPA GMTs and GMT ratios with 95% CIs were calculated using a cLDA model. Per protocol, within-group MOD were not calculated.
Time Frame: Day 30 postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Titers
  Serotype 6A | 1663.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 464.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 5030.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 807.16 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 3641.84 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1565.56 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 2459.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 244.49 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 2620.19 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 62.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 2065.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 167.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 2742.93 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 110.53 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 1699.54 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 66.24 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B | 4992.58 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 349.07 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Serotype 6A; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 3.58, 95% CI 2-sided [1.86 to 6.88] — V116/PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Serotype 15A; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 6.23, 95% CI 2-sided [3.54 to 10.98] — V116/PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Serotype 15C; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 2.33, 95% CI 2-sided [1.23 to 4.39] — V116/PNEUMOVAX™23
Statistical Analysis 4: Comparison: V116 vs PNEUMOVAX™23; Serotype 16F; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 10.06, 95% CI 2-sided [5.39 to 18.78] — V116/PNEUMOVAX™23
Statistical Analysis 5: Comparison: V116 vs PNEUMOVAX™23; Serotype 23A; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 42.09, 95% CI 2-sided [19.67 to 90.03] — V116/PNEUMOVAX™23
Statistical Analysis 6: Comparison: V116 vs PNEUMOVAX™23; Serotype 23B; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 12.37, 95% CI 2-sided [6.97 to 21.94] — V116/PNEUMOVAX™23
Statistical Analysis 7: Comparison: V116 vs PNEUMOVAX™23; Serotype 24F; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 24.82, 95% CI 2-sided [11.65 to 52.86] — V116/PNEUMOVAX™23
Statistical Analysis 8: Comparison: V116 vs PNEUMOVAX™23; Serotype 31; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 25.66, 95% CI 2-sided [14.65 to 44.93] — V116/PNEUMOVAX™23
Statistical Analysis 9: Comparison: V116 vs PNEUMOVAX™23; Serotype 35B; Test type: Other — GMT ratio and 95% CI are estimated from a cLDA model; GMT Ratio = 14.30, 95% CI 2-sided [8.72 to 23.47] — V116/PNEUMOVAX™23

7. Secondary Outcome: Serotype-specific IgG GMCs for the Unique Serotypes in V116
Description: The GMCs for serotype-specific pneumococcal IgG antibodies unique to V116 were measured using PnECL. Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% CIs were calculated using a cLDA model. Per protocol, within-group MOD were not calculated.
Time Frame: Day 30 postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
μg/mL
  Serotype 6A | 6.38 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A | 16.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.04 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C | 21.42 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.81 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F | 5.57 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.43 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A | 4.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.48 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B | 8.56 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2.06 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F | 13.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.49 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31 | 5.25 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.51 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B | 24.61 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.54 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 vs PNEUMOVAX™23; Serotype 6A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 3.00, 95% CI 2-sided [1.73 to 5.19] — V116/PNEUMOVAX™23
Statistical Analysis 2: Comparison: V116 vs PNEUMOVAX™23; Serotype 15A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 8.03, 95% CI 2-sided [4.61 to 13.98] — V116/PNEUMOVAX™23
Statistical Analysis 3: Comparison: V116 vs PNEUMOVAX™23; Serotype 15C; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 3.14, 95% CI 2-sided [1.77 to 5.58] — V116/PNEUMOVAX™23
Statistical Analysis 4: Comparison: V116 vs PNEUMOVAX™23; Serotype 16F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 13.06, 95% CI 2-sided [8.45 to 20.19] — V116/PNEUMOVAX™23
Statistical Analysis 5: Comparison: V116 vs PNEUMOVAX™23; Serotype 23A; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 8.55, 95% CI 2-sided [5.19 to 14.09] — V116/PNEUMOVAX™23
Statistical Analysis 6: Comparison: V116 vs PNEUMOVAX™23; Serotype 23B; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 4.15, 95% CI 2-sided [2.72 to 6.36] — V116/PNEUMOVAX™23
Statistical Analysis 7: Comparison: V116 vs PNEUMOVAX™23; Serotype 24F; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 28.68, 95% CI 2-sided [16.59 to 49.58] — V116/PNEUMOVAX™23
Statistical Analysis 8: Comparison: V116 vs PNEUMOVAX™23; Serotype 31; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 10.27, 95% CI 2-sided [6.71 to 15.73] — V116/PNEUMOVAX™23
Statistical Analysis 9: Comparison: V116 vs PNEUMOVAX™23; Serotype 35B; Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 15.95, 95% CI 2-sided [11.62 to 21.90] — V116/PNEUMOVAX™23

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Baseline in GMTs of Serotype-specific OPA
Description: GMTs for the serotypes in V116 and PNEUMOVAX™23 were determined using the MOPA at baseline and 30 days post vaccination and derived from a cLDA model. The GMFR (Day 30 GMT/Day 1 GMT) from baseline (Day 1) to Day 30 of each pneumococcal serotype was calculated.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: All randomized participants without deviations from the protocol that may have substantially affected the results of this immunogenicity endpoint and who had sufficient data to perform the analyses for each serotype
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Ratio
  Serotype 3 | 9.86 [7.07 to 13.75] | 6.35 [4.43 to 9.10]
  Serotype 7F: number analyzed (Participants) | 50 | 51
  Serotype 7F | 19.79 [10.60 to 36.94] | 21.53 [11.79 to 39.30]
  Serotype 19A | 10.80 [7.27 to 16.04] | 6.74 [4.45 to 10.18]
  Serotype 22F: number analyzed (Participants) | 51 | 49
  Serotype 22F | 15.14 [8.25 to 27.79] | 18.13 [9.17 to 35.85]
  Serotype 33F | 11.47 [8.20 to 16.04] | 11.62 [7.91 to 17.06]
  Serotype 8 | 102.33 [75.07 to 139.50] | 48.14 [32.69 to 70.88]
  Serotype 9N: number analyzed (Participants) | 49 | 51
  Serotype 9N | 55.49 [31.26 to 98.50] | 40.11 [22.97 to 70.03]
  Serotype 10A: number analyzed (Participants) | 49 | 49
  Serotype 10A | 31.29 [15.34 to 63.81] | 21.93 [12.29 to 39.11]
  Serotype 11A: number analyzed (Participants) | 51 | 48
  Serotype 11A | 42.06 [25.15 to 70.32] | 20.68 [12.11 to 35.33]
  Serotype 12F: number analyzed (Participants) | 48 | 50
  Serotype 12F | 94.74 [54.15 to 165.76] | 44.70 [24.59 to 81.24]
  Serotype 17F: number analyzed (Participants) | 51 | 49
  Serotype 17F | 23.63 [13.40 to 41.68] | 11.40 [7.07 to 18.40]
  Serotype 20A | 11.69 [7.27 to 18.81] | 5.94 [4.12 to 8.57]
  Serotype 6A: number analyzed (Participants) | 50 | 51
  Serotype 6A | 22.76 [12.66 to 40.93] | 8.31 [5.24 to 13.17]
  Serotype 15A | 10.70 [6.31 to 18.13] | 3.02 [1.67 to 5.43]
  Serotype 15C: number analyzed (Participants) | 50 | 48
  Serotype 15C | 36.53 [18.49 to 72.15] | 16.72 [9.39 to 29.76]
  Serotype 16F: number analyzed (Participants) | 51 | 50
  Serotype 16F | 14.74 [8.27 to 26.28] | 1.84 [1.10 to 3.06]
  Serotype 23A: number analyzed (Participants) | 50 | 51
  Serotype 23A | 46.69 [25.58 to 85.22] | 1.93 [1.05 to 3.56]
  Serotype 23B: number analyzed (Participants) | 50 | 51
  Serotype 23B | 43.21 [25.15 to 74.23] | 4.43 [3.00 to 6.54]
  Serotype 24F: number analyzed (Participants) | 47 | 45
  Serotype 24F | 9.21 [5.06 to 16.78] | 0.75 [0.40 to 1.40]
  Serotype 31 | 27.99 [16.04 to 48.85] | 1.22 [0.75 to 2.01]
  Serotype 35B | 7.39 [4.32 to 12.67] | 0.56 [0.41 to 0.78]
  Serotype 6C: number analyzed (Participants) | 51 | 50
  Serotype 6C | 5.63 [3.17 to 9.99] | 4.00 [2.21 to 7.24]
  Serotype 15B: number analyzed (Participants) | 50 | 49
  Serotype 15B | 35.68 [18.43 to 69.08] | 23.54 [13.35 to 41.50]
  Serotype 20B: number analyzed (Participants) | 49 | 49
  Serotype 20B | 6.08 [3.16 to 11.71] | 8.89 [5.29 to 14.95]

9. Secondary Outcome: GMFR From Baseline in Serotype-specific IgG GMCs
Description: GMCs for the serotypes in V116 and PNEUMOVAX™23 were measured by PnECL at baseline and 30 days post vaccination and derived from a cLDA model. The GMFR (Day 30 GMC/Day 1 GMC) from baseline (Day 1) to Day 30 of each pneumococcal serotype was calculated.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 | PNEUMOVAX™23
Number analyzed (Participants) | 51 | 51
Ratio
  Serotype 3 | 5.92 [4.25 to 8.24] | 4.47 [3.48 to 5.74]
  Serotype 7F | 23.86 [16.20 to 35.14] | 10.51 [7.57 to 14.58]
  Serotype 19A | 7.58 [5.51 to 10.44] | 3.52 [2.71 to 4.56]
  Serotype 22F | 14.68 [9.24 to 23.30] | 6.57 [4.65 to 9.28]
  Serotype 33F | 21.61 [14.49 to 32.23] | 11.52 [8.24 to 16.13]
  Serotype 8 | 31.58 [22.46 to 44.39] | 16.71 [12.61 to 22.14]
  Serotype 9N | 24.26 [16.60 to 35.46] | 10.56 [8.01 to 13.92]
  Serotype 10A | 15.70 [10.45 to 23.59] | 7.19 [5.13 to 10.07]
  Serotype 11A | 9.31 [6.51 to 13.31] | 4.64 [3.47 to 6.22]
  Serotype 12F | 23.87 [15.22 to 37.44] | 6.53 [4.52 to 9.44]
  Serotype 17F | 20.71 [15.14 to 28.33] | 7.37 [5.60 to 9.69]
  Serotype 20A | 11.68 [8.14 to 16.77] | 6.19 [4.57 to 8.38]
  Serotype 6A | 14.01 [8.99 to 21.86] | 4.67 [3.28 to 6.63]
  Serotype 15A | 32.11 [18.79 to 54.89] | 3.34 [2.52 to 4.44]
  Serotype 15C | 42.20 [25.71 to 69.25] | 11.50 [7.83 to 16.88]
  Serotype 16F | 21.00 [14.13 to 31.23] | 1.52 [1.33 to 1.73]
  Serotype 23A | 18.42 [12.28 to 27.63] | 2.26 [1.67 to 3.06]
  Serotype 23B | 14.04 [9.14 to 21.58] | 3.22 [2.55 to 4.06]
  Serotype 24F | 31.58 [18.26 to 54.60] | 1.15 [1.01 to 1.31]
  Serotype 31 | 17.97 [12.37 to 26.10] | 1.64 [1.28 to 2.09]
  Serotype 35B | 16.93 [11.99 to 23.90] | 1.10 [1.05 to 1.15]
  Serotype 6C: number analyzed (Participants) | 49 | 50
  Serotype 6C | 5.94 [4.25 to 8.30] | 2.21 [1.79 to 2.74]
  Serotype 15B | 11.14 [7.39 to 16.78] | 8.61 [6.14 to 12.08]

ADVERSE EVENTS:
Time Frame: Up to 62 days postvaccination.
Description: The analysis population for All-Cause Mortality included all randomized participants. The safety analysis population included all randomized participants who received the study vaccination.
Arm/Group | V116 | PNEUMOVAX™23
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 30/51 | 35/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 (N=51) | PNEUMOVAX™23 (N=51)
Fatigue (General disorders) | 7 (7) | 5 (5)
Injection site erythema (General disorders) | 5 (5) | 5 (5)
Injection site pain (General disorders) | 28 (28) | 34 (34)
Injection site swelling (General disorders) | 7 (7) | 7 (7)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
Headache (Nervous system disorders) | 5 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT04665050/Prot_SAP_000.pdf